CLINICAL TRIAL: NCT07158112
Title: A Randomized Three-Month Clinical Trial Evaluating Anti-Gingivitis Efficacy of Stannous Fluoride Dentifrices Relative to a Negative Control
Brief Title: Assessing Gingivitis and Plaque From a Marketed Toothpaste
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025029
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positive Control (Active Comparator): 0.454% stannous fluoride
  Interventions: Drug: Stannous Fluoride Dentifrice
- Negative Control (Active Comparator): 0.76% Sodium Monofluorophosphate
  Interventions: Drug: Sodium monofluorophosphate dentifrice
- Test Product (Active Comparator): 0.454% stannous fluoride
  Interventions: Drug: Test Stannous Fluoride Dentifrice

INTERVENTIONS:
Drug: Stannous Fluoride Dentifrice — Each subject will be randomly assigned to one of three treatment products and will be asked to brush 2x a day (1 minute per brushing) for 3 months.
  Arms: Positive Control
Drug: Test Stannous Fluoride Dentifrice — Each subject will be randomly assigned to one of three treatment products and will be asked to brush 2x a day (1 minute per brushing) for 3 months.
  Arms: Test Product
Drug: Sodium monofluorophosphate dentifrice — Each subject will be randomly assigned to one of three treatment products and will be asked to brush 2x a day (1 minute per brushing) for 3 months.
  Arms: Negative Control

SUMMARY:
The primary objective of this study is to evaluate the effect of two 0.454% stannous fluoride dentifrices on gingivitis relative to a negative control (Colgate® Cavity Protection toothpaste) and the comparative anti-gingivitis efficacy of the two 0.454% SnF2 dentifrices after 12 weeks of product use.

ELIGIBILITY:
Inclusion Criteria:

i. Be at least 18 years of age; ii. Provide consent prior to study participation and receive a signed copy of the Informed Consent form; iii. Be in good general health as determined by the Investigator/Designee based on a review of their medical history; iv. Have at least 16 gradable teeth; v. Have mild to moderate gingivitis with 10%-70% bleeding sites; vi. Agree to return for scheduled visits and follow the study procedures; vii. Agree to refrain from use of any non-study oral hygiene products for the duration of the study; viii. Agree to delay any elective dentistry, including dental prophylaxis, until the completion of the study; ix. Agree to refrain from any oral hygiene for 12 hours prior to their next visit; x. Agree to refrain from eating, drinking using tobacco in any form (including smoking substances such as marijuana, vaping products, e-cigarettes), flossing, using toothpicks, using medicated lozenges and/or breath mints, or chewing gum at least 4 hours from your next study visit (exception allowed: small sips of water up until 45 minutes prior to their appointment); and, xi. Agree not to participate in any other oral care studies for the duration of this study.

Exclusion Criteria:

i. Having taken medications (antibiotic, anti-inflammatory, or anti-coagulant) which could alter gingival bleeding within 4 weeks of the Baseline Visit; ii. Have any oral conditions that could interfere with study compliance and/or examination procedures, such as widespread caries, soft or hard tissue tumor of the oral cavity, or advanced periodontal disease; iii. Have any of the following: fixed orthodontic appliances or attachments for aligner treatment, lower bonded retainers; removable partial dentures, iv. Have a history of allergies or hypersensitivity to ingredients in commercial dental products or cosmetics; v. Had oral/gum surgery within the previous two months; vi. Nursing, self-reported pregnancy or the intention of becoming pregnant any time during the course of this study; vii. A condition requiring the need for antibiotic premedication prior to dental procedures or use within 2 weeks of the Baseline visit; or viii. Have any condition or disease, as determined by the Investigator/Designee based on a review of the medical history which could be expected to interfere with examination procedures or with the subject's safe completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2025-12-07 (Estimated); Study Completion 2025-12-07 (Estimated)

PRIMARY OUTCOMES:
Number of Bleeding Sites | 1 month and 3 months
  Number of Bleeding Sites

SECONDARY OUTCOMES:
Loe-Silness Gingival Evaluation | 1 month and 3 months
  Evaluation of bleeding and gum inflammation
Turesky Plaque Evaluation | 1 month and 3 months
  Evaluation of Plaque

CONTACTS AND LOCATIONS:
Overall Officials: Nachnani, Principal Investigator — University Health Resources Group, Inc.
Locations (1):
- University Health Resources Group, Whitter, California, United States